CLINICAL TRIAL: NCT03181464
Title: Sphenopalatine Ganglion Nerve Block for Postdural Puncture Headache in Obstetrics
Acronym: SNoB
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201703055
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Postdural Puncture Headache; Cerebrospinal Fluid Leak; Spinal; Puncture, Complications, Headache
MeSH Terms: conditions — Post-Dural Puncture Headache; Cerebrospinal Fluid Leak; Headache | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled cross-over trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental - lidocaine 4% (Experimental): Continuous infusion lidocaine at 3ml/hr for 1 hour bilaterally onto the posterior wall of the nasopharynx.
  Interventions: Drug: Lidocaine 4%
- placebo comparator (Placebo Comparator): Continuous infusion saline at 3ml/hr for 1 hour bilaterally onto the posterior wall of the nasopharynx
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine 4% — lidocaine solution
  Other Names: Xylocaine
  Arms: experimental - lidocaine 4%
Drug: Placebo — saline .9% injection
  Other Names: saline
  Arms: placebo comparator

SUMMARY:
During labor and delivery, pregnant women may choose to receive pain relief called epidural analgesia, which is the delivery of a numbing agent through the back and into a body space around the spinal column. This numbs the area of the stomach and the pelvis. Typically the numbing agent is lidocaine, which is a local anesthetic like your dentist uses. Some times the numbing agent is combined with another medication that causes drowsiness and relieves pain called a narcotic. One of the risks associated with having this kind of pain relief is unintentional puncture of a sheath of tissue that surrounds and protects the spinal cord when inserting the needle. This sheath is called the dura. This would cause the fluid surrounding the spinal cord to leak out and this would cause a headache. This headache is called a post-dural puncture headache [PDPH]. The headache can be mild or severe. Rarely, PDPH can be serious and cause bleeding or small clots in the brain and damage to nerves that come out of the brain.

The purpose of this study is to test the use of a technique that uses a hollow cotton swab [no needles] to numb a nerve cell cluster that sits at the very back of the nasal cavity. The anatomical name for this nerve cell cluster is the sphenopalatine ganglion. This has been done before at BJH and other hospitals with positive results, but no formal studies have been conducted here. Also, the sphenopalatine ganglion [SPG] has been the treatment target for other kinds of headaches. To numb the SPG, a hollow tip cotton swab [like a long Q-Tip] is inserted through the nose to the back of the nasal cavity and a solution of numbing agent is slowly pumped through the hollow Q-tip. This study will include a group that will receive a salt solution through the swab instead of a numbing agent. Subjects will be offered BJH standard care for their headache if they do not have relief from the study procedures. Standard care would be decided by their treating physician and may include oral pain medications and/or medications like ibuprofen [Motrin] or they could have a procedure called an epidural blood patch. This is performed by injecting a small amount of the patient's own blood into the areas of the spinal column where the original epidural anesthesia was injected in order to "patch" the leaks in the dura.

ELIGIBILITY:
Inclusion Criteria:

* A parturient who received an epidural or CSE for either labor or cesarean delivery - including attempted epidural; irrespective of whether a diagnosis of inadvertent spinal was noted at the time.
* A patient complaining of symptoms of postural headache consistent with postdural puncture headache. This is defined by the ICHD-II (International Classification of Headache Disorders-II) as one of the following symptoms to be present: headache, neck stiffness, tinnitus, hypoacusis (auditory deficit), photophobia, or nausea - symptoms which occur within 15 minutes of moving to an upright position (sitting or standing) and resolving within 15 minutes of moving to the supine position.

Exclusion Criteria:

* Single-shot spinal anesthesia (unless an epidural was attempted).
* Epidural performed for non-obstetric indications.
* Patient with a clinically suspected diagnosis of meningitis, intracranial hemorrhage or venous thrombosis - unless these have been excluded by neurological assessment and/or imaging as appropriate for normal clinical management.
* Symptoms or signs of cranial nerve palsy: e.g., diplopia.
* Contraindication to performance of epidural blood patch.
* Patient refusal or inability to understand consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women, 1 day postpartum
Enrollment: 0 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Subject-reported analgesia | 1 hour after infusion
  Number of subjects reporting resolution of headache

SECONDARY OUTCOMES:
Subject-reported lack of effectiveness | 1 hour after infusion
  Number of subjects reporting no impact of treatment on headache and requesting blood patch

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ginosar, MBBS, Principal Investigator — WUDA, Washington University School of Medicine
Locations (1):
- Washington University in St Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No